CLINICAL TRIAL: NCT02391259
Title: Randomized, Multicenter, Double-Blind, Placebo-Controlled, Rising Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 557 in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of AMG 557 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060132
Record Dates: First submitted 2015-01-06; First posted 2015-03-18 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — AMG 557

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 557 (Experimental): AMG 557 administered as subcutaneous and intravenous doses.
  Interventions: Drug: AMG 557
- Placebo (Placebo Comparator): No active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 557 — AMG 557 is for the treatment of sybjects with systemic lupus erythematosus
  Arms: AMG 557
Drug: Placebo — contains no active drug
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, sequential rising single-dose study in which approximately 56 subjects with SLE will be enrolled in 7 dosing cohorts

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE with positive ANA
* Stable disease with no change in SLE therapy within the previous 30 days
* BMI from 18 to 38 kg/m2

Exclusion Criteria:

* Have had signs or symptoms of a viral, bacterial or fungal infection within 30 days of study randomization
* Evidence of renal disease or liver disease
* Any history of granulomatous disease including autoimmune granulomatous vasculitis and sarcoidosis
* Prior administration of any other biologic that primarily targets the immune system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From 29 days to 169 days
  Subject incidence of treatment-emergent adverse events, vital signs, physical examinations, clinical laboratory safety tests, and ECGs

SECONDARY OUTCOMES:
Pharmacokinetic profile of AMG 557 including Tmax, AUClast and Cmax | From 29 days to 169 days
  Serum concentration and derived PK parameters including Tmax, AUClast and Cmax

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (10):
  - Research Site, Anniston, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Michigan City, Indiana
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Sullivan BA, Tsuji W, Kivitz A, Peng J, Arnold GE, Boedigheimer MJ, Chiu K, Green CL, Kaliyaperumal A, Wang C, Ferbas J, Chung JB. Inducible T-cell co-stimulator ligand (ICOSL) blockade leads to selective inhibition of anti-KLH IgG responses in subjects with systemic lupus erythematosus. Lupus Sci Med. 2016 Apr 8;3(1):e000146. doi: 10.1136/lupus-2016-000146. eCollection 2016. PMID 27099766
- [Derived] Welcher AA, Boedigheimer M, Kivitz AJ, Amoura Z, Buyon J, Rudinskaya A, Latinis K, Chiu K, Oliner KS, Damore MA, Arnold GE, Sohn W, Chirmule N, Goyal L, Banfield C, Chung JB. Blockade of interferon-gamma normalizes interferon-regulated gene expression and serum CXCL10 levels in patients with systemic lupus erythematosus. Arthritis Rheumatol. 2015 Oct;67(10):2713-22. doi: 10.1002/art.39248. PMID 26138472
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com